CLINICAL TRIAL: NCT06847542
Title: A Phase IIIb, Multicenter, Single-arm Study Assessing the Effectiveness, Safety and Patient Reported Outcomes of a 36-week Refill Exchange Regimen for the Port Delivery System With Ranibizumab in Patients With Neovascular Age-related Macular Degeneration
Brief Title: A Study of 36-Week Refill Exchanges of Port Delivery System (PDS) With Ranibizumab in nAMD
Acronym: Sightspire
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MR45625; 2024-516924-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: This is a Phase 3b study.
Masking Description: The outcome assessor (Visual acuity assessor) will be blinded.
  * The best corrected visual acuity (BCVA) examiner will only conduct refraction and BCVA assessments and will be masked to participant study eye assignment and study visit type.
  * The BCVA examiner will have no access to a participant's BCVA scores from previous visits and will be aware only of the participant's refraction data from previous visits.
  * The BCVA examiner may provide no other direct or indirect participant care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Port Delivery System (PDS) (Experimental): Participants will have the PDS implant (pre-filled with 100 mg/mL of ranibizumab) [approximately 2-milligrams (mg) dose] surgically inserted in the study eye on Day 1. Participants who meet the disease activity criteria (DAC) at Week 24 or receive supplemental treatment with intravitreal (IVT) injections of ranibizumab prior to Week 24 will receive implant refill exchanges every 24 weeks (Q24W). Participants who do not meet the DAC at Week 24 and have not received supplemental treatment will receive PDS refill exchanges Q36W.
  Interventions: Device: Susvimo PDS Implant; Drug: Ranibizumab

INTERVENTIONS:
Device: Susvimo PDS Implant — Ranizumab will be administered via a PDS implant per the schedule described in the arm.
  Other Names: RO4893594
Drug: Ranibizumab — Participants will receive ranibizumab delivered through the PDS implant.
  Participants will receive ranibizumab, 0.5 mg IVT injections as a supplemental treatment.
  Other Names: RO4893594

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety, and PROs of the port delivery system with ranibizumab 100 milligrams/milliliters (mg/mL) refilled every 36 weeks (Q36W) in participants with nAMD.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of nAMD within 24 months prior to screening
* Previous treatment with at least 3 anti-vascular endothelial growth factor (VEGF) IVT injections for nAMD per standard of care within 6 months prior to screening
* Demonstrated response to prior anti-VEGF IVT treatment since diagnosis
* Availability of historical VA data obtained at or after nAMD diagnosis and prior to the first anti-VEGF treatment for nAMD
* Availability of historical OCT image data obtained at or after nAMD diagnosis and prior to the first anti-VEGF treatment for nAMD
* BCVA of 34 letters or better using ETDRS chart at a starting distance of 4 meters at screening and enrollment visits

Exclusion Criteria:

A. Prior Ocular Treatment

Study Eye:

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for age-related macular degeneration (AMD)
* Previous treatment with corticosteroid intravitreal injection
* Previous intraocular device implantation
* History of vitreous hemorrhage
* History of rhegmatogenous retinal detachment
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery
* History of corneal transplant

Either Eye:

* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the ranibizumab injections, study-related procedure preparations (including fluorescein), dilating drops, or any of the anesthetic and antimicrobial preparations used by a participant during the study
* Prior participation in a clinical trial involving any experimental therapies for nAMD
* Prior treatment with brolucizumab or gene therapy for nAMD

B. Macular Neovascularization/Choroidal Neovascularization (MNV/CNV) Lesion Characteristics:

Study Eye:

* Subretinal hemorrhage that involves the center of the fovea
* Subfoveal fibrosis or subfoveal atrophy

Either Eye:

* CNV due to other causes, such as ocular histoplasmosis, trauma, central serous chorioretinopathy, or pathologic myopia
* CNV masquerading lesions

C. Concurrent Ocular Conditions:

Study Eye:

* Subfoveal and/or juxtafoveal retinal pigment epithelial tear
* Any concurrent intraocular condition that would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results
* Active intraocular inflammation
* Retinal tears or peripheral retinal breaks on depressed fundus exam that are untreated or treated within 3 months prior to the enrollment visit
* Aphakia or absence of the posterior capsule
* Uncontrolled ocular hypertension or glaucoma
* History or presence of severe posterior blepharitis, recurrent chalazia or hordeolum, severe dry eye syndrome, or severe allergic conjunctivitis
* Trichiasis
* Corneal neuropathy
* Lagophthalmos or incomplete blink
* Active or history of facial nerve palsy/paresis

Fellow (Non-study) Eye:

- Non-functioning non-study eye defined as either: BCVA of hand motion or worse OR no physical presence of non-study eye (i.e., monocular)

Either Eye:

* Any active or history of uveitis
* Active or history of keratitis, scleritis, endophthalmitis, or chronic blepharitis
* Suspected or active ocular or periocular infectious conjunctivitis or endophthalmitis
* Active or history of floppy eyelid syndrome
* Active thyroid eye disease

D. Concurrent Systemic Conditions:

* Uncontrolled blood pressure
* Active or history of autoimmune diseases
* History of stroke within the last 3 months prior to informed consent
* Atrial fibrillation diagnosed or worsened within the last 3 months prior to informed consent
* History of myocardial infarction (MI) within the last 3 months prior to informed consent
* Confirmed active systemic infection
* History of other disease, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab or placement of the implant and that might affect interpretation of the results of the study
* Use of any systemic anti-VEGF agents
* Chronic use of oral corticosteroids
* Active cancer within 12 months of enrollment except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2028-09-12 (Estimated); Study Completion 2028-10-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Best Corrected Visual Acuity (BCVA) Score Averaged Over Weeks 68 and 72, as Assessed Using the Early Treatment Diabetic Retinopathy Study (ETDRS) Chart at a Starting Distance of 4 Meters | Baseline, Week 68, Week 72
  BCVA letters were measured using EDTRS chart while participants were at a starting distance of 4 meter. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in visual acuity (VA).

SECONDARY OUTCOMES:
Change From Baseline in BCVA Score Over Time | From baseline up to Week 72
  BCVA letters were measured using EDTRS chart while participants were at a starting distance of 4 meter. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.
Percentage of Participants Who Lose ≤ 15, ≤ 10, ≤ 5, or Gain ≥ 0 Letters in BCVA Score From Baseline Over Time | From baseline up to Week 72
  BCVA letters were measured using EDTRS chart while participants were at a starting distance of 4 meter. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.
Change From Baseline in Center Point Thickness (CPT) | From baseline up to Week 72
Change From Baseline in Central Subfield Thickness (CST) | From baseline up to Week 72
Proportion of Participants Who do not Undergo Supplemental Treatment With IVT Ranibizumab Before Each Refill-exchange Procedure | Up to Week 72
Number of Supplemental Treatments Participants Received in Each Refill Cycle | Up to Week 72
Frequency of Study Visits in Each Refill Cycle | Up to Week 72
Proportion of Participants Who Report Preferring PDS Compared With IVT Ranibizumab Treatment as Measured by the PDS Patient Preference Questionnaire (PPPQ) at Weeks 24 and 72 | Weeks 24 and 72
Proportion of Participants With Bilateral Disease Who Report Preferring PDS Compared With IVT Ranibizumab Treatment Measured by the PPPQ at Weeks 24 and 72 | Weeks 24 and 72
Number of Participants With Ocular and Systemic (Non-ocular) Adverse Events (AEs) | Up to approximately 19 months
Number of Participants With Adverse Events of Special Interests (AESIs) and their Severity, Including Ocular AESIs | Up to approximately 19 months
Number of Participants With Ocular AESIs and Severity of Ocular AESIs During the Post-operative and Follow-up Period | Post-operative period: ≤ 37 days of initial implantation surgery Follow-up period: > 37 days after implantation surgery (up to 72 weeks)
Number of Participants With Adverse Device Effects (ADEs) and Severity of ADEs With PDS | Up to approximately 19 months
Number of Participants With Anticipated Serious Adverse Device Effects (ASADEs) and Severity of ASADEs With PDS | Up to approximately 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Kepler Universitätskliniken GmbH - Med Campus III, Linz
  - Landesklinikum Mistelbach, Mistelbach
- Klaudianova Nemocnice - Mlada Boleslav;Ophtalmology dpt, Mladá Boleslav, Czechia
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark
- France (5):
  - Institut Ophtalmologique De l Ouest Jules Verne, Nantes, Paris
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - Clinique Honore Cave, Montauban
  - CHNO des Quinze Vingts, Paris
  - CHU Poitiers - CHR La Miletrie, Poitiers
- Medizinische Hochschule Hannover, Klinik für Augenheilkunde, Hanover, Germany
- Greece (4):
  - "G.Gennimatas" General Hospital of Athens, Athens, Attica
  - Attikon University General Hospital, Chaïdári
  - University General Hospital of Heraklion, Heraklon
  - University Hospital of Larissa, Larissa
- Italy (2):
  - Ospedale Monaldi - AORN dei Colli, Napoli, Campania
  - Ospedale Isola Tiberina - Gemelli Isola;UOC Chirurgia Vitreoretinica, Rome, Lazio
- Poland (5):
  - MW-med, Krakow, Lesser Poland Voivodeship
  - Klinika Okulistyczna ?Jasne Blonia? Sp. z o. o., ?ód?
  - Szpital sw. Lukasza, Bielsko-Bia?a
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
- South Korea (6):
  - Kyungpook National University Hospital, Daegu
  - Ajou University Medical Center, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Switzerland (2):
  - Berner Augenklinik, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Maharaj Nakorn ChiangMai Hospital, Chiang Mai
- United Kingdom (2):
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Moorfields Eye Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing